CLINICAL TRIAL: NCT02543736
Title: Reliability and Validity of Gait and Postural Balance Parameters Using an Instrumented Treadmill in Patients With Knee Osteoarthritis
Brief Title: Reliability and Validity of Gait and Postural Balance Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Treadmill Study
Record Dates: First submitted 2015-08-28; First posted 2015-09-07 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- Instrumented Treadmill System (Other): The Instrumented Treadmill System records vertical ground reaction force and pressures.
  Interventions: Device: Instrumented Treadmill System

INTERVENTIONS:
Device: Instrumented Treadmill System — Patients will perform twice a gait and a balance analysis on an instrumented treadmill system combined to a photoelectric cell system while controls will only perform once.
  Other Names: Photoelectric Cell System

SUMMARY:
Knee osteoarthritis (KOA) patients, have impairments in gait and balance. Accurate gait and postural balance analysis is needed to detect this impairments. Nevertheless methodological quality about the recording of gait and balance analysis in KOA patients is lacking in literature.

DETAILED DESCRIPTION:
In patients with knee osteoarthritis (KOA), impairments in gait and balance are well recognized and therefore objective and accurate gait and postural balance analysis is crucial to detect potential alterations in balance and gait function in this patient group.

Gait analysis in orthopaedic patients has been mainly investigated during level walking at a self-selected speed or at pre-determined gait velocities. Nevertheless, walking at a comfortable speed may not necessary result in any gait impairments and therefore the use of more challenging tasks is probably required. In addition, some patients are not able to walk at a required walking speed or slope, because of pain and disability. Therefore it seems reasonable to evaluate gait parameters of KOA patients while walking at different speeds and surface inclinations.

Postural balance parameters are also important outcome measures in the assessment of KOA patients. Postural stability is generally assessed throughout the quantification of the displacement and velocity of the centre of pressure (COP) with larger excursions and higher velocities indicating poorer balance.

Recently, instrumented treadmill systems (ITS) have been introduced for the evaluation of spatiotemporal and kinetic gait as well as postural balance parameters throughout a capacitance-based foot pressure platform. Further, they permit an assessment of the gait parameters at different speeds and slopes. Spatiotemporal and kinetic gait parameters provided by ITS have been shown to be valid and reliable during level walking in healthy young and elderly persons and during walking at different speeds and slopes. ITS can also be used for the quantification of static balance, because they are able to provide the velocity and displacement changes of COP. However the validity and reliability of gait and postural balance analysis at different slopes and speeds in patients with KOA are lacking.

Similarly to ITS, photoelectric cell systems (PCS) also permit the quantification of spatiotemporal gait parameters but in addition they are portable, their set up is very quick, they are relatively cheap and can be adapted to a treadmill. PCS have been shown to be both valid and reliable for the assessment of spatiotemporal gait parameters in healthy adults and also in KOA patients.

The main aim of this study is to evaluate the methodological quality of postural and gait parameters assessed at different treadmill inclinations and velocities using an ITS in patients with KOA. In particular, we will investigate the test-retests reliability, the discriminant validity and the concurrent validity.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 85 years.
* Men and women.
* Unilateral symptomatic KOA.
* Patient in waitlist at the Schulthess Clinic for knee arthroplasty.
* Living place: Canton of Zurich or neighbouring Cantons.
* Signed written informed consent.

Exclusion Criteria:

* Symptomatic OA in lower extremity joints other than the knee.
* Bilateral symptomatic KOA.
* Usage of walking aids.
* Surgery to the lower limbs in the prior 12 months.
* BMI >35 kg/m2.
* Disorders that affect gait or balance function.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Spatial gait Parameter: step length (cm) | baseline
Temporal gait Parameter: cadence (step/min) | baseline
Postural Balance Parameter: Centre of pressure path length (cm) | baseline
Postural Balance Parameter: Centre of pressure velocity (m/s) | baseline

SECONDARY OUTCOMES:
Spatial gait Parameter: step width (cm) | baseline
Temporal gait Parameter: single limb support (% of gait cycle) | baseline
Kinetic gait Parameter: heel/toe force (N) | baseline
Postural Balance Parameter: Centre of pressure displacement in the medio-lateral and antero-posterior direction (mm) | baseline
Postural Balance Parameter: Centre of pressure area (mm2) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Casartelli, PhD, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

REFERENCES:
- [Background] Bejek Z, Paroczai R, Illyes A, Kiss RM. The influence of walking speed on gait parameters in healthy people and in patients with osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2006 Jul;14(7):612-22. doi: 10.1007/s00167-005-0005-6. Epub 2005 Dec 6. PMID 16331521
- [Background] Elbaz A, Mor A, Segal G, Debi R, Shazar N, Herman A. Novel classification of knee osteoarthritis severity based on spatiotemporal gait analysis. Osteoarthritis Cartilage. 2014 Mar;22(3):457-63. doi: 10.1016/j.joca.2013.12.015. Epub 2014 Jan 10. PMID 24418677
- [Background] Faude O, Donath L, Roth R, Fricker L, Zahner L. Reliability of gait parameters during treadmill walking in community-dwelling healthy seniors. Gait Posture. 2012 Jul;36(3):444-8. doi: 10.1016/j.gaitpost.2012.04.003. Epub 2012 May 1. PMID 22555061
- [Background] Hinman RS, Bennell KL, Metcalf BR, Crossley KM. Balance impairments in individuals with symptomatic knee osteoarthritis: a comparison with matched controls using clinical tests. Rheumatology (Oxford). 2002 Dec;41(12):1388-94. doi: 10.1093/rheumatology/41.12.1388. PMID 12468818
- [Background] Lee M, Song C, Lee K, Shin D, Shin S. Agreement between the spatio-temporal gait parameters from treadmill-based photoelectric cell and the instrumented treadmill system in healthy young adults and stroke patients. Med Sci Monit. 2014 Jul 14;20:1210-9. doi: 10.12659/MSM.890658. PMID 25017613
- [Background] Lee MM, Song CH, Lee KJ, Jung SW, Shin DC, Shin SH. Concurrent Validity and Test-retest Reliability of the OPTOGait Photoelectric Cell System for the Assessment of Spatio-temporal Parameters of the Gait of Young Adults. J Phys Ther Sci. 2014 Jan;26(1):81-5. doi: 10.1589/jpts.26.81. Epub 2014 Feb 6. PMID 24567681
- [Background] Lienhard K, Schneider D, Maffiuletti NA. Validity of the Optogait photoelectric system for the assessment of spatiotemporal gait parameters. Med Eng Phys. 2013 Apr;35(4):500-4. doi: 10.1016/j.medengphy.2012.06.015. Epub 2012 Jul 18. PMID 22818403
- [Background] Reed LF, Urry SR, Wearing SC. Reliability of spatiotemporal and kinetic gait parameters determined by a new instrumented treadmill system. BMC Musculoskelet Disord. 2013 Aug 21;14:249. doi: 10.1186/1471-2474-14-249. PMID 23964707
- [Background] Sorensen RR, Jorgensen MG, Rasmussen S, Skou ST. Impaired postural balance in the morning in patients with knee osteoarthritis. Gait Posture. 2014 Apr;39(4):1040-4. doi: 10.1016/j.gaitpost.2014.01.002. Epub 2014 Jan 8. PMID 24480548
- [Background] Zeni JA Jr, Higginson JS. Differences in gait parameters between healthy subjects and persons with moderate and severe knee osteoarthritis: a result of altered walking speed? Clin Biomech (Bristol). 2009 May;24(4):372-8. doi: 10.1016/j.clinbiomech.2009.02.001. Epub 2009 Mar 13. PMID 19285768
- [Background] Hassan BS, Mockett S, Doherty M. Static postural sway, proprioception, and maximal voluntary quadriceps contraction in patients with knee osteoarthritis and normal control subjects. Ann Rheum Dis. 2001 Jun;60(6):612-8. doi: 10.1136/ard.60.6.612. PMID 11350851
- [Background] Duffell LD, Southgate DF, Gulati V, McGregor AH. Balance and gait adaptations in patients with early knee osteoarthritis. Gait Posture. 2014 Apr;39(4):1057-61. doi: 10.1016/j.gaitpost.2014.01.005. Epub 2014 Jan 19. PMID 24582072
- [Background] Mills K, Hunt MA, Ferber R. Biomechanical deviations during level walking associated with knee osteoarthritis: a systematic review and meta-analysis. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1643-65. doi: 10.1002/acr.22015. PMID 23554153
- [Background] Turcot K, Hagemeister N, de Guise JA, Aissaoui R. Evaluation of unipodal stance in knee osteoarthritis patients using knee accelerations and center of pressure. Osteoarthritis Cartilage. 2011 Mar;19(3):281-6. doi: 10.1016/j.joca.2010.12.007. Epub 2010 Dec 22. PMID 21184837